CLINICAL TRIAL: NCT05074394
Title: A Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Intranasal STI-2099 (COVI-DROPS™) as Treatment for COVID-19 Infection in Outpatient Adults
Brief Title: Randomized Study to Evaluate Intranasal Dose of STI-2099 (COVI-DROPS™) in Outpatient Adults With Mild COVID-19 Infection
Acronym: US
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: to be replaced with a different protocol
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRP-COV-206US
Record Dates: First submitted 2021-10-07; First posted 2021-10-12 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: COVID19; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — STI-2020

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-DROPS (Experimental): 40 mg of COVI-DROPS administered intranasally
  Interventions: Biological: COVI-DROPS
- Placebo (Placebo Comparator): 2 mL placebo administered intranasally
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: COVI-DROPS — COVI-DROPS is a fully human monoclonal antibody that is a neutralizing antibody to SARS-CoV-2
  Other Names: STI-2099
  Arms: COVI-DROPS
Drug: Placebo — Diluent solution
  Arms: Placebo

SUMMARY:
This is prospective double-blind study in the United States is designed to investigate the efficacy and safety of a single dose of COVI-DROPS or matched placebo in outpatient adults with mild symptoms associated with COVID-19 and a recent positive COVID-19 test.

DETAILED DESCRIPTION:
Subjects will be randomized 2:1 to receive a single dose of COVI-DROPS (40 mg) or placebo in a double-blind manner. Investigational product (COVI-DROP or placebo) will be administered once on Study Day 1 and followed to Day 29. Subjects will be stratified based upon prior history of infection or vaccination versus the group who is unvaccinated and not previously infected with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Positive for COVID-19 with any approved RT-PCR or rapid antigen test within 7 days of planned treatment
* Have mild illness/symptoms based upon NIH criteria. The NIH illness severity definition for "mild" states as follows: "Individuals who have any of the various signs and symptoms of COVID-19 (e.g., fever, cough, sore throat, malaise, headache, muscle pain, nausea, vomiting, diarrhea, loss of taste and smell) but who do not have shortness of breath, dyspnea, or abnormal chest imaging."
* Be in good health as judged by investigator using screening medical history and physical examination. Participants who are otherwise healthy with a stable chronic medical condition may enroll
* A prior COVID-19 infection in the past from which the subject fully recovered or a previously unknown asymptomatic infection is allowed, as is any previous COVID-19 vaccination
* Must be willing and able to comply with all planned study procedures and be available for all study visits and follow-up as required by the protocol
* Subject must have provided written informed consent which includes signing the institutional review board or independent ethics committee approved consent form prior to participating in any study related activity
* Willing to follow contraception guidelines

Exclusion Criteria:

* In the investigator's opinion, has moderate or severe symptoms or rapidly progressive symptoms which are likely to progress such that a hospitalization is imminent (within 24-48 hours)
* Currently using chronic oxygen therapy due to an underlying comorbidity and requires an increase in baseline oxygen flow rate due to COVID-19 infection
* Is an immunocompromised subject even if previously fully vaccinated against COVID-19 or recovered from a prior COVID-19 infection
* Has an active documented infection other than COVID-19
* Any medical condition that, in the Investigator's opinion, could adversely impact safety or key objectives of the study, particularly any intranasal pathology or disease process
* Pregnant or lactating women who are breast feeding or planning on either during the study
* Has received within the 30 days prior to screening or is planning on receiving an EUA-cleared monoclonal antibody (mAb) during the study
* Has participated or is participating in a clinical research study evaluating COVID-19 convalescent plasma, other non-EUA-cleared mAbs against COVID-19 or intravenous immunoglobulin within 3 months or less than 5 half-lives of the investigational product (whichever is longer) prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who have a COVID-19-related visit or hospitalization | Baseline through Day 29
  Proportion of subjects with COVID-19-related urgent medically attended visits, emergency department assessments, hospitalizations ≥ 24h or all-cause death through Day 29 (D29)

SECONDARY OUTCOMES:
Viral load change from baseline to Day 15 (D15) | Baseline through Day 15
  Viral load change from baseline to D15 based on nasal quantitative reverse transcription polymerase chain reaction (RT-PCR) COVID-19 viral titers (Log-10 copies/mL). Includes viral load change for subjects in the unvaccinated/no prior infection group as well as the vaccinated/prior infection group
Proportion of subjects who have a COVID-19-related visit or hospitalization based on stratification groups | Baseline to Day 29
  For each of the unvaccinated/no prior infection group or the vaccinated/prior infection group, proportion of subjects with COVID-19-related urgent medically attended visits, emergency department assessments, hospitalizations ≥ 24h or all-cause death through D29

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.